CLINICAL TRIAL: NCT02873026
Title: A Phase 3 Multi-centre Double-masked Randomised Controlled Trial of Adjunctive Intraocular and Periocular Steroid (Triamcinolone Acetonide) Versus Standard Treatment in Eyes Undergoing Vitreoretinal Surgery for Open Globe Trauma.
Brief Title: Adjunctive Steroid Combination in Ocular Trauma (ASCOT) Study
Acronym: ASCOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHAD1031
Record Dates: First submitted 2016-06-13; First posted 2016-08-19 (Estimated); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Eye Injury Trauma
MeSH Terms: interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (No Intervention): The patient will receive the standard care given to all patients that have received a vitrectomy following open globe trauma.
- Triamcinolone acetonide (Experimental): Triamcinolone Acetonide 4mg/0.1ml intravitreal cavity and 40mg/1ml subtenons to be injected at the time of the vitrectomy. Patients will then receive standard care following operation.
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide — Following the repair of the open globe eye trauma, the use of Triamcinolone Acetonide will be investigated
  Other Names: kenalog
  Arms: Triamcinolone acetonide

SUMMARY:
Eye trauma is a leading cause of blindness and visual impairment. Penetrating injuries of the eye are more likely to result in poor vision and the main cause of this is a scarring response on the retina (proliferative vitreoretinopathy, PVR) The purpose of this study is to investigate the potential of an anti-inflammatory treatment (triamcinolone acetonide) to improve the outcome of surgery in eyes that have suffered severe trauma.There is good evidence from laboratory studies that additional steroid treatment into and around the eye at the time of surgery could reduce scarring by reducing inflammation and improve visual outcomes.

DETAILED DESCRIPTION:
Trauma is an important cause of visual impairment and blindness worldwide and a leading cause of blindness in young adult males.Globally it has been estimated that 1.6 million people are blind as a result of ocular trauma with 2.3 million suffering bilateral low vision. Ocular trauma is the commonest cause of unilateral blindness in the world today with up to 19 million with unilateral blindness or low vision. It is estimated that almost one million people in the United States live with trauma-related visual impairment. Ocular trauma has extensive socio-economic costs - patients with open globe injuries lose a mean of 70 days of work. In the United States work related eye injuries cost over $300 million per year (www.prevent blindness.org) this equates to an annual cost to the UK economy (for which no comparable data exists) of £37.5 million.

In the UK it is estimated that 5000 patients per year sustain eye injuries serious enough to require hospital admission and of these 250 will be permanently blinded in the injured eye. Recent European studies document incidences of 2.4 and 3.2 per 100000 per year for open-globe injuries which suggests an annual incidence for the UK of between 1500 and 2000.

Ocular injuries which result in visual loss invariably affect the posterior segment of the eye and prevention of visual loss involves posterior segment (vitreoretinal) surgery. It is clear from recent published data that although vitreoretinal surgical techniques have improved, outcomes remain unsatisfactory and that development of the intraocular scarring response proliferative vitreoretinopathy (PVR) is the leading cause of this.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects (Aged 18 years or over at the time of enrolment)
2. Full thickness, open-globe ocular trauma undergoing vitrectomy
3. Ability to give written informed consent
4. Willingness to accept randomization and attend follow-up for 6 months.

Exclusion Criteria:

1. Children (Age less than 18 years old at time of enrollment)
2. Pre-existing uncontrolled uveitis - Patients with pre-existing uveitis are likely to be rare in the study population however they have a pre-disposition to a more aggressive form of proliferative vitreoretinopathy and will therefore be excluded. (This does not include patients whose uveitis is secondary to their injury or retinal detachment)
3. Definitive diagnosis of previous steroid induced glaucoma - these patients are at risk of steroid related pressure rise and will be excluded (this does not include patients in whom a query of previous steroid-induced raised IOP has been postulated)
4. Pregnant or Breastfeeding females (Females of childbearing potential must be willing to use an effective method of contraception (hormonal or barrier method of birth control; true abstinence) from the time consent is signed until 6 weeks after their completion of the trial. Females of childbearing potential must have a negative urinary pregnancy test within 7 days prior to being registered for trial treatment (Subjects are considered not of child bearing potential if they are permanently sterile (i.e. they have undergone a hysterectomy, bilateral tubal occlusion, or bilateral salpingectomy) or they are postmenopausal)
5. Allergy or previous known adverse reaction to triamcinolone acetonide
6. Inability to attend regular follow up
7. Unable to give written informed consent
8. Current or planned systemic corticosteroid use of a dose above physiological levels (e.g. >10mg prednisolone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Improvement of visual acuity at 6 months | 6 months
  The proportion of patients with an improvement from baseline to 6 months of at least 10 on the corrected visual acuity in the study eye (total ETDRS letter score measured at 4 metres and 1 metre)

SECONDARY OUTCOMES:
Total visual acuity score at 6 months | 6 months
  Total EDTRS score in the study eye at the 6 months follow up appointment

CONTACTS AND LOCATIONS:
Overall Officials: David Charteris, MD, Principal Investigator — Moorfields Eye Hosptial
Locations (1):
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ezeofor V', Anthony BF, Bryning L, Casswell EJ, Cro S, Cornelius VR, Bunce C, Robertson E, Kelly J, Murphy C, Banerjee PJ, Charteris DG, Edwards RT. Economic evaluation of an adjunctive intraocular and peri-ocular steroid vitreoretinal surgery for open globe trauma: Cost-effectiveness of the ASCOT randomised controlled trial. PLoS One. 2024 Dec 16;19(12):e0311158. doi: 10.1371/journal.pone.0311158. eCollection 2024. PMID 39680515
- [Derived] Casswell EJ, Cro S, Cornelius VR, Banerjee PJ, Zvobgo TM, Tudor Edwards R, Ezeofor V, Anthony B, Shahid SM, Bunce C, Kelly J, Murphy C, Robertson E, Charteris D; ASCOT Investigator Study Group. Randomised controlled trial of adjunctive triamcinolone acetonide in eyes undergoing vitreoretinal surgery following open globe trauma: The ASCOT study. Br J Ophthalmol. 2024 Feb 21;108(3):440-448. doi: 10.1136/bjo-2022-322787. PMID 36849205